CLINICAL TRIAL: NCT02598544
Title: Atrial Natriuretic Peptide (ANP)-Induced Lipid Mobilization Regulation in Different Adipose Tissue Depots of Obese Subjects
Brief Title: Endocrine Regulation of Lipolysis in Obesity and Diabetes
Acronym: ERLO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Dominique Hansen, prof. dr., Hasselt University
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 14.17/REVA14.02
Record Dates: First submitted 2015-10-16; First posted 2015-11-06 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Obesity; Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- lean men (Other)
  Interventions: Other: adipose tissue sampling
- Obese men without type 2 diabetes (Other)
  Interventions: Other: adipose tissue sampling
- Obese men with type 2 diabetes (Other)
  Interventions: Other: adipose tissue sampling

INTERVENTIONS:
Other: adipose tissue sampling — adipose tissue (subcutaneous and visceral adipose tissue) sampling during abdominal surgery and phenotype determination

SUMMARY:
Adipose tissue (AT) dysfunction is a commonly observed feature of metabolic dysfunction in obesity and diabetes. An important characteristic when examining AT function is the capacity to break down stored lipids (i.e. lipolysis) and its regulation. In the present study, the aim was to investigate whether atrial natriuretic peptide-mediated lipolysis is altered in different adipose tissue depots (subcutaneous and visceral adipose tissue) of obese subjects with or without type 2 diabetes, compared to age-matched lean men. Eventually, the knowledge gained from this research will contribute to a better understanding of the present adipose tissue dysfunction and to the optimization of exercise programs for people with obesity and diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Lean group: BMI < 25 kg/m², insulin sensitive (HOMA-Insuline Resistance (IR) < 2.3), age 40-65
* Obese groups: BMI > 30 kg/m², presence or absence of type 2 diabetes based on use of glucose lowering medication or HbA1c > 6.5%, age 40-65

Exclusion Criteria:

* presence of a history of heart, lung or kidney disease and/or presence of endocrine anomalies. Use of beta-blockade medication.

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2013-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Glycerol release by mature adipocytes, isolated from subcutaneous and visceral adipose tissue, upon stimulation with isoprenalin or ANP (ex vivo) | day 1
  Investigation of concentration effect of ISO/ANP on lipolysis (glycerol release) by mature adipocytes isolated from adipose tissue biopsies, glycerol release is measured in the incubation medium following a 3 hour incubation period. Measured for adipose tissue (subcutaneous and visceral adipose tissue) of both lean and obese subjects
ANP receptor expression profiles on mRNA and protein level in both adipose tissue depots for both lean and obese subjects. | day 1
  Receptor expression determination in order to clarify the underlying mechanism responsible for possible differences in lipolytic responses.
Adipose tissue inflammation | day 1
  Adipose tissue inflammation (by means of FACS analysis) and its relation to insulin sensitivity and adipose tissue function in lean, obese and obese diabetics subjects.

SECONDARY OUTCOMES:
Body composition | day 1
  Body composition (body fath percentage), measured by BIA
BMI (kg/m²) | day 1
body height (m) | day 1
weight (kg) | day 1
hip circumference (cm) | Day 1
waist (cm) | Day 1
blood glucose | day 1
blood insuline | day 1
blood FFA | day 1
blood triglycerides | day 1
blood glycated hemoglobin | day 1
blood ANP | day 1
  fasting blood sample to determine blood glucose, insulin, FFA, , glycated hemoglobin and ANP
blood pressure (mmHg) | Day 1
Concomitant medication | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Hansen, prof. dr., Principal Investigator — Hasselt University; Ellen Blaak, prof. dr., Principal Investigator — Maastricht University; Kenneth Verboven, drs., Study Chair — Hasselt University
Locations (4):
- Belgium (3):
  - Hasselt University, Diepenbeek
  - Ziekenhuis Oost-Limburg, Genk
  - Jessa Ziekenhuis, Hasselt
- Maastricht University, Maastricht, Netherlands